CLINICAL TRIAL: NCT01806753
Title: Performance of Endoscopic Submucosal Dissection According to the Sedation Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2012-0661
Record Dates: First submitted 2013-03-05; First posted 2013-03-07 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Early Gastric Cancer; Gastric Adenoma
Keywords: Endoscopic submucosal dissection; Sedation; Propofol; Midazolam
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- midazolam/propofol injection (Experimental): Intermittent midazolam/propofol injection controlled by endoscopist
  Interventions: Procedure: Intermittent midazolam/propofol injection controlled by endoscopist
- propofol infusion (Active Comparator): Continuous propofol infusion with opioid administration
  Interventions: Procedure: Continuous propofol infusion with opioid administration

INTERVENTIONS:
Procedure: Intermittent midazolam/propofol injection controlled by endoscopist — In this arm1, sedation during endoscopic submucosal dissection is controlled by endoscopists.
  First, pethidine 50 mg with midazolam 0.05 mg/kg are injected in a bolus fashion.
  When the patient seems to be discomfort or the patient's movements were observed, endoscopists should check the Modified Observer Assessment of Alertness/Sedation (MOAAS).
  If MOAAS is 5 or 6, propofol 0.25 mg/kg will be injected. Otherwise, pethidine 12.5 mg will be injected.
  Arms: midazolam/propofol injection
Procedure: Continuous propofol infusion with opioid administration — In this arm2, sedation during endoscopic submucosal dissection is controlled by anesthesiologists.
  First, remifentanil 0.5 ug/kg with propofol 0.5 mg/kg are injected in a bolus fashion.
  Then, remifentanil 0.08 ug/kg/min and propofol 2 mg/kg/h are infused continuously.
  When the patient seems to be discomfort or the patient's movements were observed, anesthesiologists should check the MOAAS.
  If MOAAS is 5 or 6, infusion rate of propofol will be increased by 0.5 mg/kg/h. Otherwise, infusion rate of remifentanil will be increased by 0.02 ug/kg/min.
  Arms: propofol infusion

SUMMARY:
Although proper sedation is mandatory for endoscopic procedures such as endoscopic submucosal dissection, the effects of sedation on ESD performance and complications have not been fully evaluated. In the investigators previous retrospective study, en bloc resection and complete resection rates, and procedure time could be improved by sedation with continuous propofol infusion with opioid administration by anesthesiologists. However, there are several limitations to the study including retrospective design. The investigators aimed to evaluate the relationship among sedation methods, satisfaction of endoscopists or patients, clinical outcomes, and complications after endoscopic submucosal dissection for gastric neoplasia.

ELIGIBILITY:
Inclusion Criteria:

1. Age, between 20 and 80
2. Early gastric cancer or adenoma, which is indicated by endoscopic submucosal dissection
3. ECOG performance status 0 or 1
4. American Society of Anesthesiologist Physical Status 1, 2, or 3

Exclusion Criteria:

1. Previous subtotal gastrectomy
2. Previous gastrostomy
3. Repeated endoscopic submucosal dissection
4. Three or more synchronous lesions
5. Allergy to midazolam, propofol, fentanyl, or remifentanil
6. Pregnancy or breast milk feeding
7. Active infection
8. Significant cardiopulmonary disease
9. Active hepatitis or severe hepatic dysfunction
10. Severe renal dysfunction
11. Severe bone marrow dysfunction
12. Severe neurologic or psychotic disorder

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2013-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Satisfaction of endoscopists | Within 10 minutes from the end of the endoscopic submucosal dissection

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Park CH, Shin S, Lee SK, Lee H, Lee YC, Park JC, Yoo YC. Assessing the stability and safety of procedure during endoscopic submucosal dissection according to sedation methods: a randomized trial. PLoS One. 2015 Mar 24;10(3):e0120529. doi: 10.1371/journal.pone.0120529. eCollection 2015. PMID 25803441